CLINICAL TRIAL: NCT06988631
Title: Investigation of the Effect of Foot Sole Sensory Training on Sensorimotor Organization in Individuals With General Joint Hypermobility
Brief Title: Sensorimotor Organization in Individuals With General Joint Hypermobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Principal Investigator, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16/07/28.12.2023
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Generalized Joint Hypermobility
Keywords: joint hypermobility; food sense; Sensorimotor
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kontrol group (Active Comparator): Participants were given brochures and training on foot care and health.
  Interventions: Other: foot care booklet
- exercise group (Experimental): Participants were asked to practice the foot sole sensory training program at home every day for 2 weeks.
  Interventions: Other: Sensory treatment

INTERVENTIONS:
Other: Sensory treatment — Participants were asked to practice the foot sole sensory training program at home every day for 2 weeks.
  Arms: exercise group
Other: foot care booklet — Participants were given a booklet about healthy feet and were informed.
  Arms: Kontrol group

SUMMARY:
This study is the first to examine the effect of sole sensory training on sensorimotor organization in individuals with GEH. Individuals with a Beighton score of 5 and above were included in the study. Within the scope of the study, individuals with general joint hypermobility (GEH) were divided into intervention and control groups by the Randomization method. The intervention group received sole sensory training in the home environment. Both groups were given a foot care brochure. The individuals' sole sensory and balance skills were evaluated before and after the intervention. As a result of the study, the intervention aimed to prevent injuries and disabilities that may occur due to joint laxity by improving sole sensory and balance.

ELIGIBILITY:
Inclusion Criteria:

* Persons with a Beighton score ≥5 without any systemic disease
* Asymptomatic persons

Exclusion Criteria:

* People who have had an upper or lower extremity injury in the last 3 months,
* People who have a history of fractures or surgery in the last year,
* People who have been pregnant in the last year,
* Those diagnosed with Ehlers-Danlos Syndrome (EDS), hypermobile Ehlers-Danlos syndrome (hEDS), or hypermobility spectrum disorders (HSD)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Light touch sensation | 2 weeks
  It was evaluated using the Semmes-Weinstein Monofilament (SWM) test kit.
Two-Point Separation sensation | 2 weeks
  A discriminator was used to assess two-point discrimination perception.
Vibration sense | 2 weeks
  A 128 Hz tuning fork was used to evaluate vibration sensation.

SECONDARY OUTCOMES:
Proprioception | 2 weeks
  Joint position sense test for proprioception assessment was performed using a digital goniometer device.
Muscle Strength | 2 weeks
  A hand-held dynamometer (Lafayette Instrument®, Layafette, IN) was used to determine muscle strength for both lower extremities of the individuals.
Balance | 2 weeks
  Dynamic balance of individuals was assessed with the Y Balance Test.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum technical university, Erzurum, State/Province, Turkey (Türkiye)